CLINICAL TRIAL: NCT04181463
Title: Inhalation Approaches to Nausea: A Randomized Controlled Trial
Brief Title: Nasal Inhalation of Isopropyl Alcohol for the Treatment of Nausea in Patients With Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0472; NCI-2019-07377 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0472 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-11-19; First posted 2019-11-29 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — 2-Propanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (isopropyl alcohol) (Experimental): Patients receive isopropyl alcohol via nasal inhalation.
  Interventions: Drug: Isopropyl Alcohol; Other: Questionnaire Administration
- Arm II (placebo) (Placebo Comparator): Patients receive placebo via nasal inhalation.
  Interventions: Other: Placebo; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Isopropyl Alcohol — Given via nasal inhalation
  Other Names: Isopropanol; Isopropanolol
  Arms: Arm I (isopropyl alcohol)
Other: Placebo — Given via nasal inhalation
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
The goal of this research study is to understand the effect of inhalation approaches in reducing nausea in cancer patients.

DETAILED DESCRIPTION:
In this study, inhalation of a study solution will be compared to inhalation of placebo, both in the form of preparation pads (a small square of material that contains the solution). Isopropyl alcohol may be a part of the preparation pads. A placebo is not a drug. It looks like the study solution but is not designed to treat any disease or illness. It is designed to be compared with the study solution to learn if the study solution has any real effect.

Inhalation of the study solution may help to control your nausea. Future patients may benefit from what is learned. There may be no benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including side effects, potential expenses, and time commitment.

ELIGIBILITY:
Inclusion Criteria:

* Rate current severity of acute/chronic nausea >= 4 on NRS (Numeric Rating Scale)
* Diagnosis of cancer
* Able to read/write in English
* Referred to supportive care service as an inpatient or outpatient
* Rate anxiety as =< 4 on ESAS-FS (Edmonton Symptom Assessment Scale-Financial Distress and Spiritual Pain)
* Participants must agree to inhale isopropyl alcohol

Exclusion Criteria:

* Received anti-emetics in the last 30 minutes
* Received medical procedures (e.g. blood draws) which required exposure of isopropyl alcohol in the last 30 minutes
* Inability to inhale through nares (including recent upper respiratory infection)
* Known allergy to isopropyl alcohol
* Delirium (i.e., score >= 7 on the Memorial Delirium Assessment Scale [MDAS])
* Have never been on anti-emetics during the course of the treatment here (anti-emetic naive)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-11-05 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in nausea | Baseline up to 5 minutes post-intervention
  The mean change in nausea level will be compared between the two arms by two sample t-test. In case there's any violation in the underlying assumptions (e.g. normality, equality of variance, etc.) proper transformation (e.g. logarithm, square root, etc.) or non-parametric methods (Wilcoxon rank sum test) will be applied.

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne J Heung, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org